CLINICAL TRIAL: NCT06138990
Title: Pharmacoscopy-guided Clinical Standard-of-care in Relapsed/Refractory Acute Myeloid Leukemia, a Randomized Phase-2 Clinical Trial
Brief Title: Pharmacoscopy-guided Clinical Standard-of-care in r/r AML
Acronym: RAPID-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ETH Zurich (Other)
Collaborators: University of Zurich (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RAPID-01
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-09

CONDITIONS: AML, Adult
Keywords: relapsed / refractory AML; Pharmacoscopy; Functional precision medicine
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: This is a randomised, controlled, parallel group, superiority interventional trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm: Pharmacoscopy-guided clinical standard-of-care (Experimental): Patients in the PCY-guided treatment arm will receive one of the clinical standard-of-care treatments suggested by their own PCY results, and confirmed by the treating physician.
  Interventions: Diagnostic Test: Pharmacoscopy
- Control arm (Active Comparator): Patients in the control arm will be treated with clinical standard-of-care therapy for RR AML selected by the physician (physician's choice).
  Interventions: Drug: Clinical standard-of-care (physician's choice)

INTERVENTIONS:
Diagnostic Test: Pharmacoscopy — Pharmacoscopy (PCY) is an image-based ex vivo drug testing platform developed by the Snijder lab at the ETH Zurich. PCY measures in the drug response of patient cells from small biopsies using automated microscopy and single-cell image analysis. PCY prioritizes treatments based on their specific efficacy against AML cells, while minimizing toxicity to healthy (non-malignant) cells in the patient biopsy.
  Arms: Intervention arm: Pharmacoscopy-guided clinical standard-of-care
Drug: Clinical standard-of-care (physician's choice) — Clinical standard-of-care therapy for RR AML selected by the physician (physician's choice).
  Arms: Control arm

SUMMARY:
With an overall survival of below 12 months, the outcome of relapsed/refractory AML (RR AML) is poor, making it a critical challenge to identify effective therapies at this stage. The RAPID-01 trial aims to show for the first time in a randomized and controlled clinical trial that Pharmacoscopy (PCY), a functional precision medicine platform, helps improve clinical standard-of-care treatment selection for patients suffering from relapsed/refractory AML.

ELIGIBILITY:
Inclusion criteria

* Patient with refractory or relapsed AML according to ELN2022 criteria.
* Age 18-70 years.
* Considered to be eligible for intensive chemotherapy.
* Written informed consent.

Exclusion criteria

* Acute promyelocytic leukemia (APL) with PML-RARA or one of the other pathognomonic variant fusion genes/chromosome translocations.
* Blast crisis after chronic myeloid leukemia (CML).
* Considered not eligible for intensive chemotherapy.
* Condition of the patient does not allow to wait for PCY results (patient requires immediate treatment).
* PCY not working / patient sample did not pass the QC steps of PCY.
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the principal investigator may interfere with the project or affect patient compliance.
* Legal incompetence or Subjects lacking capacity to provide informed consent.
* Participation in a clinical trial with an investigational drug within the 30 days preceding and during the present investigation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate at day 28 | day 28

SECONDARY OUTCOMES:
Composite response rate (CR+CRh+CRi) at day 28 | day 28
Rate of patients bridged to allogeneic hematopoietic stem cell transplantation within 3 months post-treatment initiation | 3 months
Treatment-related mortality within 3 months post-treatment initiation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Theocharides, MD PhD, Principal Investigator — University of Zurich
Locations (2):
- Switzerland (2):
  - Inselspital Bern, Bern, Canton of Bern
  - University Hospital Zurich, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data will be made available upon publication of the study results in a peer-reviewed internationally recognized journal.
Supporting Information: CSR
Time Frame: De-identified patient data will be made available upon publication of the study results in a peer-reviewed internationally recognized journal.

REFERENCES:
- [Background] Snijder B, Vladimer GI, Krall N, Miura K, Schmolke AS, Kornauth C, Lopez de la Fuente O, Choi HS, van der Kouwe E, Gultekin S, Kazianka L, Bigenzahn JW, Hoermann G, Prutsch N, Merkel O, Ringler A, Sabler M, Jeryczynski G, Mayerhoefer ME, Simonitsch-Klupp I, Ocko K, Felberbauer F, Mullauer L, Prager GW, Korkmaz B, Kenner L, Sperr WR, Kralovics R, Gisslinger H, Valent P, Kubicek S, Jager U, Staber PB, Superti-Furga G. Image-based ex-vivo drug screening for patients with aggressive haematological malignancies: interim results from a single-arm, open-label, pilot study. Lancet Haematol. 2017 Dec;4(12):e595-e606. doi: 10.1016/S2352-3026(17)30208-9. Epub 2017 Nov 15. PMID 29153976
- [Background] Kornauth C, Pemovska T, Vladimer GI, Bayer G, Bergmann M, Eder S, Eichner R, Erl M, Esterbauer H, Exner R, Felsleitner-Hauer V, Forte M, Gaiger A, Geissler K, Greinix HT, Gstottner W, Hacker M, Hartmann BL, Hauswirth AW, Heinemann T, Heintel D, Hoda MA, Hopfinger G, Jaeger U, Kazianka L, Kenner L, Kiesewetter B, Krall N, Krajnik G, Kubicek S, Le T, Lubowitzki S, Mayerhoefer ME, Menschel E, Merkel O, Miura K, Mullauer L, Neumeister P, Noesslinger T, Ocko K, Ohler L, Panny M, Pichler A, Porpaczy E, Prager GW, Raderer M, Ristl R, Ruckser R, Salamon J, Schiefer AI, Schmolke AS, Schwarzinger I, Selzer E, Sillaber C, Skrabs C, Sperr WR, Srndic I, Thalhammer R, Valent P, van der Kouwe E, Vanura K, Vogt S, Waldstein C, Wolf D, Zielinski CC, Zojer N, Simonitsch-Klupp I, Superti-Furga G, Snijder B, Staber PB. Functional Precision Medicine Provides Clinical Benefit in Advanced Aggressive Hematologic Cancers and Identifies Exceptional Responders. Cancer Discov. 2022 Feb;12(2):372-387. doi: 10.1158/2159-8290.CD-21-0538. Epub 2021 Oct 11. PMID 34635570
- [Background] Schmid JA, Festl Y, Severin Y, Bacher U, Kronig MN, Snijder B, Pabst T. Efficacy and feasibility of pharmacoscopy-guided treatment for acute myeloid leukemia patients who have exhausted all registered therapeutic options. Haematologica. 2024 Feb 1;109(2):617-621. doi: 10.3324/haematol.2023.283224. No abstract available. PMID 37439341
- See also: Snijder Lab website — https://www.snijderlab.org